CLINICAL TRIAL: NCT02666950
Title: A Phase 2 Study of WEE1 Inhibition With AZD1775 Alone or Combined With Cytarabine in Patients With Advanced Acute Myeloid Leukemia and Myelodysplastic Syndrome
Brief Title: WEE1 Inhibitor AZD1775 With or Without Cytarabine in Treating Patients With Advanced Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1488; NCI-2015-02136 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1488 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2016-01-08; First posted 2016-01-28 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2018-11

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome With Isolated Del(5q); Myelodysplastic/Myeloproliferative Neoplasm; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Chromosome 5q Deletion Syndrome; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute | interventions — Cytarabine; adavosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm B (cytarabine and WEE1 inhibitor AZD1775 (Experimental): Patients receive cytarabine and WEE1 inhibitor AZD1775 as in Arm A.
  Interventions: Drug: Cytarabine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: WEE1 Inhibitor AZD1775
- Arm C (WEE inhibitor AZD1775) (Experimental): Patients receive WEE inhibitor AZD1775 PO daily on days 1-5, 8-12, 15-19, and 22-26.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: WEE1 Inhibitor AZD1775

INTERVENTIONS:
Drug: Cytarabine — Given SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm B (cytarabine and WEE1 inhibitor AZD1775
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: WEE1 Inhibitor AZD1775 — Given PO
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775

SUMMARY:
This randomized phase II trial studies how well WEE1 inhibitor AZD1775 with or without cytarabine works in treating patients with acute myeloid leukemia or myelodysplastic syndrome that has spread to other places in the body and usually cannot be cured or controlled with treatment. WEE1 inhibitor AZD1775 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving WEE1 inhibitor AZD1775 works better with or without cytarabine in treating patients with advanced acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the clinical efficacy of AZD1775 (WEE1 inhibitor AZD1775) in combination with AraC (cytarabine) in patients with newly diagnosed acute myeloid leukemia (AML) by assessing complete response (complete remission [CR] plus CR with incomplete blood count recovery [CRi]) rates.

II. To estimate the clinical efficacy of AZD1775 alone or in combination with AraC in patients with relapsed/refractory AML and hypomethylating agent failure myelodysplastic syndrome (MDS) by assessing complete response (CR plus CRi) rates.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of AZD1775 alone or combined with AraC in the study population.

II. To estimate additional measures of clinical benefit (i.e. hematological improvements, transfusion requirements).

III. To measure the duration of response of AZD1775 alone or combined with AraC.

IV. To measure time to response of AZD1775 alone or combined with AraC. V. To measure time to progression of AZD1775 alone or combined with AraC. VI. To measure overall survival of AZD1775 alone or combined with AraC. VII. To measure time to AML (for MDS subjects) of AZD1775 alone or combined with AraC.

TERTIARY OBJECTIVES:

I. To determine the pharmacokinetics (PK) of AZD1775 alone or combined with AraC in the study population.

II. To conduct correlative research studies characterizing underlying molecular events and solidifying putative mechanism of action in vivo and to identify potential pharmacodynamic/biomarkers of response to AZD1775 alone or combined with AraC.

III. To evaluate quality of life (QOL) and patient-reported symptoms in subjects treated with AZD1775 alone or combined with AraC.

OUTLINE: Elderly newly diagnosed patients are assigned to arm A.

ARM A (ELDERLY NEWLY DIAGNOSED PATIENTS): Patients receive cytarabine subcutaneously (SC) twice daily (BID) on days 1-5 and 8-12 and WEE inhibitor AZD1775 orally (PO) daily on days 1-5 and 8-12.

Patients are randomized to 1 of 2 treatment arms.

ARM B: Patients receive cytarabine and WEE1 inhibitor AZD1775 as in Arm A.

ARM C: Patients receive WEE inhibitor AZD1775 PO daily on days 1-5, 8-12, 15-19, and 22-26.

In all arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient population (histological or cytologically confirmed diagnosis):

  * Untreated elderly (> 60 years) AML if in the intermediate and poor-risk cytogenetic group and not candidates (as judged by treating doctor of medicine [MD]) for or willing to undergo standard induction therapy (i.e. elderly unfavorable cytogenetic AML) or any untreated AML age > 65 years

    * Note: previous therapy with a hypomethylating agent (HMA) for a diagnosis of MDS is allowed
  * Relapsed or refractory AML (>= 18 years)
  * Any MDS (>= 18 years) having failed or been intolerant to prior hypomethylating agent (HMA) treatment

    * Failure is defined as any disease progression while on HMA, relapse after HMA treatment or no response after 4 cycles of 5-Azacitidine or decitabine
    * Patients with isolated 5q-/5q- syndrome must have failed, not tolerated, or lenalidomide in addition to having failed or been intolerant to HMA treatment

      * Note: patients with chronic myelomonocytic leukemia (CMML) and MDS/myeloproliferative neoplasms (MPN) overlap are allowed if meeting other study eligibility criteria
      * Note: for all patient groups, therapy as part of a plan as a bridge to transplant is allowed
* Total bilirubin =< 1.5 mg/dL (except Gilbert's syndrome or known hemolysis or leukemic infiltration)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x upper limit normal (ULN) or < 5 x ULN if organ involvement
* Alkaline phosphatase < 5 x ULN
* Serum creatinine =< 2 x ULN or 24 hour creatinine (Cr) clearance > 30 ml/min
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Ability to provide informed written consent and be able to adhere to the study visit schedule and other protocol requirements
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide blood and bone marrow aspirate samples for correlative research purposes
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Men and women must be willing to use appropriate contraception throughout study and for 6 months after
* Male patients who are sexually active with a female partner of childbearing potential must be either surgically sterilized or agree to use barrier contraception (ie, condoms) for the duration of study participation, and for 90 days after the final dose of study drug; cessation of birth control after this point should be discussed with a responsible physician
* Patients who have undergone stem cell transplantation (SCT), autologous or allogeneic, are eligible provided that they are > 60 days from stem cell infusion, have graft-versus-host disease (GVHD) =< grade 1 and are off immunosuppressive agents for > 28 days at time of registration

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection, known positive for active infectious hepatitis, type A, B or C (past infection allowed), or psychiatric illness/social situations that would limit compliance with study requirements; Note: ongoing infection controlled on antibiotics/antifungal/antiviral medications are allowed
* Any of the following prior therapies:

  * Cytotoxic chemotherapy =<14 days prior to registration
  * Immunotherapy =< 14 days prior to registration
  * Biologic therapy (i.e. antibody therapies) =< 14 days prior to registration
  * Radiation therapy =<14 days prior to registration
  * Targeted therapies (i.e. kinase inhibitors, =< 7 days or 5 half-life's whichever is shorter)

    • For steroids or other non-cytotoxics given for blast count control, patient must be off for > 24 hours (hrs) before starting therapy; NOTE: hydroxyurea (HU) is allowed for blast count control throughout study
  * Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm =< 14 days prior to registration
* Active uncontrolled central nervous system (CNS) leukemia; NOTE: positive (cyto)pathology is allowed and patient can receive intrathecal chemotherapy
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Any previous treatment with AZD1775 or allergic reactions to excipients of AZD1775
* Acute promyelocytic leukemia (APL, M3) unless failed regimens that included tretinoin, arsenic trioxide, anthracyclines and cytarabine and currently NOT candidates for stem cell transplantation
* Major surgery =< 28 days prior to registration
* Clinically significant heart disease, including the following:

  * Active severe angina pectoris within 3 months prior to registration
  * Acute myocardial infarction within 3 months prior to registration
  * New York Heart Association classification IV cardiovascular disease or symptomatic class III disease

    * Note: patients with any of the above may be allowed after discussion amongst the investigators including the principal investigator
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Subject has had prescription or non-prescription drugs or other products known to be sensitive cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued two weeks prior (alternatively 5 half lives if T1/2 is known) prior to day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug

  * NOTE: co-administration of aprepitant or fosaprepitant during this study is prohibited
  * Note: individual drugs exerting CYP interactions may be continued on a case by case basis if felt essential for patient management, after discussions and discretion of the treating physician
  * The preferred azole anti-fungal medication is fluconazole (alternatively posaconazole) which can be given during treatment with AZD1775 at the treating physician's discretion, however with dose reductions of AZD1775 by 25-75% (i.e. from AZD1775 200mg to 150 or 100mg)
* Patients may not be on an inhibitor of breast cancer resistance protein (BCRP)

  * NOTE: AZD1775 is an inhibitor of breast cancer resistance protein (BCRP); the use of statins including atorvastatin which are substrates for BCRP are therefore prohibited and patients should be moved on to non-BCRP alternatives
* Not willing to avoid grapefruit, grapefruit juices, grapefruit hybrids, Seville oranges, pummelos, and exotic citrus fruits from 7 days prior to the dose of study medication and during the entire study; NOTE: orange juice is allowed
* Corrected QT interval (QTc) > 470 msec (as calculated per institutional standards) at study entry or congenital long QT syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Tibes, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients were accrued. Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm.
Groups:
- Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only): Patients receive 20 mg cytarabine (AraC) SC twice daily and 200 mg WEE1 inhibitor (AZD1775) PO daily on days 1-5 and days 8-12 OR receive only 200 mg WEE inhibitor (AZD1775) PO daily on days 1-5, 8-12, 15-19, and 22-26.
Period: Overall Study
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm.
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 1
    2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CR or CRi) Per the National Comprehensive Cancer Network (NCCN) Guidelines or According to Specific Criteria From Expert Panels
Description: Complete response rate will be evaluated over all courses of study treatment. The proportion of CR/CRi responses will be estimated by the number of CR/CRi responses divided by the total number of evaluable patients.
Time Frame: Up to 17 months
Population: Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm.
Measure: Number; unit: percentage of patients
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Number analyzed (Participants) | 3
percentage of patients | 0

2. Secondary Outcome: Clinical Benefit as Measured by the Number of Patients Who Were Not RBC Transfusion-dependent Post-Baseline
Description: Clinical benefit as measured by the number of patients who did not receive a RBC transfusion post-Baseline
Time Frame: Up to 17 months
Population: Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Duration of Response
Description: Duration of response defined for all evaluable patients who have achieved a response as the date at which the patient's earliest best objective status is first noted to be a CR/CRi response to the earliest date progression is documented
Time Frame: Up to 17 months
Population: No patients responded, thus no patients were analyzed for this outcome measure. Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm.
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Events Considered At Least Possibly Related to Treatment
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 30 days post-treatment
Population: Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm.
Measure: Number; unit: percentage of patients
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Number analyzed (Participants) | 3
percentage of patients | 100

5. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to death due to any cause.
Time Frame: From registration to death due to any cause, assessed up to 17 months
Population: Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Number analyzed (Participants) | 3
months | 6 [4.6 to 7.0]

6. Secondary Outcome: Time to Progression, Defined as the Time From Registration to the Earliest Date of Documentation of Disease Progression
Description: Time to progression (TTP) is defined to be the length of time from study registration to a) date of disease progression as defined by section 11.0 of the protocol, or b) last follow-up. If a patient dies without documentation of disease progression, the patient will be considered to have had a tumor progression at the time of death unless there is sufficient documented evidence to conclude no progression occurred prior to death. Time to progression curves were compared via the log-rank test. Progression is defined as a >25% increase in product of perpendicular diameters of contrast enhancement or mass or appearance of new lesions or unequivocal increase in size of contrast enhancement or increase in mass effect as agreed upon independently by primary physician and quality control physicians: appearance of new lesions compared to pretreatment MRI and/or CT scan.
Time Frame: Up to 17 months
Population: Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Number analyzed (Participants) | 3
months | 3.9 [3.8 to 6.9]

7. Secondary Outcome: Time to Response, Defined as the Time From Registration to the Earliest Date of Documentation of Response
Description: Time to response, defined as the time from registration to the earliest date of documentation of response. The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 17 months
Population: as for outcome 3
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Change in Biomarker Levels
Description: Continuous biomarker levels will be explored in a graphical manner including mean plots and plots of change and percent change from baseline and other summary measures. Any potential relationships between the baseline level or change in the level of each biomarker and clinical outcome such as overall response, 6-month progression and survival, and adverse event incidence will be further analyzed using Wilcoxon rank sum tests or logistic regression methods, as appropriate. Association between a dichotomized biomarker and overall response will be assessed using a chi-squared test.
Time Frame: Baseline to up to 113 days (after course 4)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Patients' Reported Outcomes as Assessed by the Brief Fatigue Inventory (BFI)
Description: BFI, as well as linear analog scales capturing early satiety, abdominal discomfort, inactivity, concentration problems, numbness/tingling in the hands/feet, night sweats, itching, bone pain, fever, and weight loss will be used.
Time Frame: Baseline to 2 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in QOL as Assessed by the European Organization for Treatment and Research of Cancer Quality of Life Questionnaire Core Questionnaire 30
Description: Scale score trajectories over time and changes from baseline over time will be examined using repeated measures or growth curve models, as appropriate, stream plots and mean plots with standard deviation error bars overall. Scores and changes at each cycle will be statistically tested using paired t-tests, and standardized response means (i.e. effect sizes) (mean of the change from baseline scores at a given cycle, divided by the standard deviation of the change scores) will be interpreted (after applying Middel's adjustment) using Cohen's cut-offs.
Time Frame: Baseline to 2 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters AUC of WEE1 Inhibitor AZD1775
Description: PK will be primarily descriptive.
Time Frame: Day 1, course 1; pre-treatment, 30 min, 1 hr, 2 hr, 4 hr, 6hr and 24 hr after WEE1 inhibitor AZD administration
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters Vd of WEE1 Inhibitor AZD1775
Description: PK will be primarily descriptive.
Time Frame: Day 1, course 1; pre-treatment, 30 min, 1 hr, 2 hr, 4 hr, 6hr and 24 hr after WEE1 inhibitor AZD administration
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters Cmax of WEE1 Inhibitor AZD1775
Description: PK will be primarily descriptive
Time Frame: Day 1, course 1; pre-treatment, 30 min, 1 hr, 2 hr, 4 hr, 6hr and 24 hr after WEE1 inhibitor AZD administration
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters Tmax of WEE1 Inhibitor AZD1775
Description: PK will be primarily descriptive
Time Frame: Day 1, course 1; pre-treatment, 30 min, 1 hr, 2 hr, 4 hr, 6hr and 24 hr after WEE1 inhibitor AZD administration
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters t1/2 of WEE1 Inhibitor AZD1775
Description: PK will be primarily descriptive
Time Frame: Day 1, course 1; pre-treatment, 30 min, 1 hr, 2 hr, 4 hr, 6hr and 24 hr after WEE1 inhibitor AZD administration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 days post-treatment
Description: Since only one patient was accrued on one arm, patient confidentiality prevents the reporting of results by arm. Each CTCAE term is a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only)
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only) (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A + Arm C (AZD1775 Combined With AraC OR AZD1775 Only) (N=3)
Anemia (Blood and lymphatic system disorders) | 3 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 3 (6)
Fever (General disorders) | 2 (3)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 3 (7)
Platelet count decreased (Investigations) | 3 (7)
White blood cell decreased (Investigations) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT02666950/Prot_SAP_000.pdf